CLINICAL TRIAL: NCT05878704
Title: A Phase I, Open-Label, Single-Dose, Non-Randomized, Parallel Group Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of GBT021601, an Oral Hemoglobin S Polymerization Inhibitor, in Adult Participants With Renal Impairment
Brief Title: Study of GBT021601 in Participants With Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision to terminate the trial after the completion of Part 1: Cohort 1 (severe renal impairment). The decision to terminate the trial was not due to any potential safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBT021601-014; C5351007 (Other: Alias Study Number)
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Renal Impairment
Keywords: End stage renal disease; Sickle Cell Disease
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): GBT021601
  Interventions: Drug: GBT021601

INTERVENTIONS:
Drug: GBT021601 — Oral

SUMMARY:
Renal Impairment study of GBT021601.

DETAILED DESCRIPTION:
This is a Phase 1, two-part, non-randomized, open-label, parallel group study to evaluate the PK, safety, and tolerability of GBT021601 following a single dose administration in adult participants with RI.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age at the time of Screening.
* Have liver (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and total bilirubin [direct and indirect]) and renal function tests, Hb, and hematocrit values within normal limits or are not clinically significant at Screening and Day -1 (Cohort 2 only).
* Has a stable renal function with no clinically significant change in renal status at least 1 month prior to study drug administration.

Exclusion Criteria:

* Any clinically significant medical history or abnormal findings upon physical examination, or clinical laboratory tests unrelated to their medical condition related to renal impairment, that might confound the results of the study or pose an additional risk in administering study drug to the participant.
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic seasonal allergies at the time of study drug administration), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease unrelated to renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Concentration of GBT021601 in whole blood and plasma | Up to 112 Days
  To evaluate the single-dose whole blood and plasma PK of GBT021601 in participants with renal impairment (RI)
Single-dose PK parameters | Up to 112 Days
  To evaluate the single-dose whole blood and plasma PK of GBT021601 in participants with renal impairment

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), clinically significant changes in laboratory assessments, electrocardiograms (ECGs), and vital signs | Up to 112 Days
  To evaluate the safety and tolerability of single dose GBT021601 in participants with renal impairment
Incidence of treatment-emergent adverse events (TEAEs), clinically significant changes in laboratory assessments, electrocardiograms (ECGs), and vital signs | Up to 112 Days
  To evaluate the safety and tolerability of GBT021601 in ESRD participants receiving IHD following a single dose

OTHER OUTCOMES:
Single-dose PK parameters for GBT021601 in RBC | Up to 112 Days
  To evaluate the single-dose RBC PK of GBT021601 in participants with RI
Amount of GBT021601 excreted in urine | Up to 112 Days
  To evaluate the urinary excretion of GBT021601 in participants with RI following a single dose
Descriptive analysis of eGFR versus PK exposure parameters | Up to 112 Days
  The relationship of eGFR, as estimated using serum creatinine and serum cystatin C on GBT021601 PK exposure in participants with RI
Protein binding of GBT021601 in plasma | Up to 112 Days
  To evaluate the protein binding of GBT021601 in participants with RI
Single-dose PK parameters for GBT021601 in RBC | Up to 112 Days
  To evaluate the single-dose RBC PK of GBT021601 in participants with ESRD receiving IHD
Extraction ratio of GBT021601 via dialysis and concentration of GBT021601 in dialysate | Up to 112 Days
  To evaluate the clearance of GBT021601 by IHD in participants with ESRD

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Orange County Research Center, Tustin, California
  - Advanced Pharma CR, LLC, Miami, Florida
  - Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-014